CLINICAL TRIAL: NCT06782022
Title: A Combination of Pre-screening for DPD Deficiency by Genotyping/phenotyping Methods and Pharmacokinetics-guided Dosing of 5-FU for Precision Treatment to Prevent Severe Toxicity in Gastrointestinal Cancer Patients.
Brief Title: DPD Guided 5-FU Precision Treatment in Gastro-intestinal Cancer Patients
Acronym: COMBIGaPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jan Gerard Maring (Other)
Responsible Party: Sponsor-Investigator, Jan Gerard Maring, PharmD, PhD (Hospital Pharmacist - Clinical Pharmacologist), Isala
Organization: Isala (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL70778.075.19
Record Dates: First submitted 2025-01-07; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Cancers
Keywords: dihydropyrimidine dehydrogenase; 5-fluorouracil; genotyping; phenotyping; therapeutic drug monitoring; fluoropyrimidines
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is designed as a single-centre prospective inception cohort study. Study duration per subject will be a maximum 3 months.
  All gastrointestinal cancer patients scheduled to treatment with fluoropyrimidine based chemotherapy will be asked to participate for the study. All patients will be screened for DPD deficiency by DPYD genotyping. Only 4 most common DPYD variants will be included, including E412E (c.1236G>A; rs56038477), I560S (*13; c.1679T>G; rs55886062), D949V (c.2846A>T; rs67376798) and IVS14 ds+1G>A (*2A; c.1905+1G>A; rs3918290). Patients will be separated into two groups: DPYD variants and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group E, DPYD wild type controls (Other): Patients without common DPYD variant will be used for this study as a control group. Patients will receive the first 5-FU-dose based on their body surface area. 5-FU plasma concentrations will be measured during cycle 1. If patients experience CTC grade 3-4 toxicity, DPYD sequencing will be performed. Dose reduction or discontinuation of 5-FU therapy will be considered according to the physician's discretion.
  Interventions: Drug: 5-Fluoro-Uracil
- Group A, DPYD E412E (c.1236G>A; rs56038477) heterozygotes (Experimental): Patients will receive the first dose based on their body surface area and gene activity score according to Clinical Pharmacogenetics Implementation Consortium (CPIC) guideline or according to the physician's descretion. Patients' blood sample will be collected once at least 4 hour after the start of the perfusion in the morning between 8 and 10 a.m. 5-FU dose for the next cycle will be calculated according to a modified algorithm of Goirand or according to the pharmacist's discretion. 5-FU plasma concentrations will be monitored until a steady state AUC of 20-30 mg.h/L is reached or a maximum 4 treatment cycles has been reached. If patients experience CTC grade 3-4 toxicity, DPYD sequencing will be performed. Dose reduction or discontinuation of 5-FU therapy will be considered according to the physician's discretion.
  Interventions: Drug: 5-Fluoro-Uracil
- Group B, DPYD IVS14 ds+1G>A (*2A; c.1905+1G>A; rs3918290) heterozygotes (Experimental): Patients will receive the first dose based on their body surface area and gene activity score according to Clinical Pharmacogenetics Implementation Consortium (CPIC) guideline or according to the physician's descretion. Patients' blood sample will be collected once at least 4 hour after the start of the perfusion in the morning between 8 and 10 a.m. 5-FU dose for the next cycle will be calculated according to a modified algorithm of Goirand or according to the pharmacist's discretion. 5-FU plasma concentrations will be monitored until a steady state AUC of 20-30 mg.h/L is reached or a maximum 4 treatment cycles has been reached. If patients experience CTC grade 3-4 toxicity, DPYD sequencing will be performed. Dose reduction or discontinuation of 5-FU therapy will be considered according to the physician's discretion.
  Interventions: Drug: 5-Fluoro-Uracil
- Group C, DPYD D949V (c.2846A>T; rs67376798) heterozygotes (Experimental): Patients will receive the first dose based on their body surface area and gene activity score according to Clinical Pharmacogenetics Implementation Consortium (CPIC) guideline or according to the physician's descretion. Patients' blood sample will be collected once at least 4 hour after the start of the perfusion in the morning between 8 and 10 a.m. 5-FU dose for the next cycle will be calculated according to a modified algorithm of Goirand or according to the pharmacist's discretion. 5-FU plasma concentrations will be monitored until a steady state AUC of 20-30 mg.h/L is reached or a maximum 4 treatment cycles has been reached. If patients experience CTC grade 3-4 toxicity, DPYD sequencing will be performed. Dose reduction or discontinuation of 5-FU therapy will be considered according to the physician's discretion.
  Interventions: Drug: 5-Fluoro-Uracil
- Group D, DPYD I560S (*13; c.1679T>G; rs55886062) heterozygotes (Experimental): Patients will receive the first dose based on their body surface area and gene activity score according to Clinical Pharmacogenetics Implementation Consortium (CPIC) guideline or according to the physician's descretion. Patients' blood sample will be collected once at least 4 hour after the start of the perfusion in the morning between 8 and 10 a.m. 5-FU dose for the next cycle will be calculated according to a modified algorithm of Goirand or according to the pharmacist's discretion. 5-FU plasma concentrations will be monitored until a steady state AUC of 20-30 mg.h/L is reached or a maximum 4 treatment cycles has been reached. If patients experience CTC grade 3-4 toxicity, DPYD sequencing will be performed. Dose reduction or discontinuation of 5-FU therapy will be considered according to the physician's discretion.
  Interventions: Drug: 5-Fluoro-Uracil

INTERVENTIONS:
Drug: 5-Fluoro-Uracil — Patients without common DPYD variant will be used for this study as a control group. Patients will receive the first 5-FU-dose based on their body surface area. 5-FU plasma concentrations will be measured during cycle 1. If patients experience CTC grade 3-4 toxicity, DPYD sequencing will be performed. Dose reduction or discontinuation of 5-FU therapy will be considered according to the physician's discretion.
  Patients with a DPYD variant will receive the first dose based on their body surface area and gene activity score according to Clinical Pharmacogenetics Implementation Consortium (CPIC) guideline or according to the physician's descretion. Patients' blood sample will be collected and the 5-FU dose for the next cycle will be calculated according to a modified algorithm of Goirand or according to the pharmacist's discretion. 5-FU plasma concentrations will be monitored until a steady state AUC of 20-30 mg.h/L is reached.

SUMMARY:
Rationale:

Fluorouracil (5-FU) are broadly used in chemotherapeutic regimens for the treatment of cancers. Dihydropyrimidine dehydrogenase (DPD) is a major enzyme in the 5-FU metabolism pathway. Patients with a partial or complete DPD deficiency have a strongly reduced capacity to metabolize 5-FU which may result in severe or life-threatening toxicity when treated with a standard dose of fluoropyrimidines. A partial DPD deficiency is present in 3-5% of the North American and European population. DPD deficiency is most often caused by genetic variants in the gene encoding DPD (DPYD). The four DPYD variants considered most clinically relevant and with statistically significant association with severe toxicity are DPYD*2A (rs3918290, c.1905+1G>A, IVS14+1G>A), c.2846A>T (rs67376798, D949V), c.1679T>G (rs55886062, DPYD*13, I560S), and c.1236G>A (rs56038477, E412E, in haplotype B3). Prospective testing for DPD deficiency can prevent severe toxicity or mortality. Several methods have been proposed for detection of DPD deficiency, based on either genotyping of DPYD or measurement of the DPD phenotype. However, DPD deficiency is not the only factor associated with variable concentrations of 5-FU. 5-FU displays an exposure-response relationship between systemic exposure and clinical events. Therapeutic Drug Monitoring (TDM) or pharmacokinetics (PK)-guided dosing of 5-FU is also considered as an alternative to ensure an acceptable exposure of 5-FU. Upfront DPD screening combined with PK guided 5-FU dosing as a tool to personalize treatment has never been studied before. In this study, we aim to investigate the PK of 5-FU for the 4 most common DPYD genetic variants, in order to better define a safe starting dose for 5-FU in DPD deficient patients.

Objectives:

The primary objective of this study is to investigate the clearance of 5-FU for the 4 most common DPYD gene variants compared to the clearance of 5-FU in DPYD wild-type patients. The secondary objectives of this study are to determine the toxicity incidence and the extent of DPD deficiency as measured by Uracil Loading Test (ULT) for the 4 most common DPYD variants, to evaluate the safety and tolerability of reduced starting dose of 5-FU in patients with DPD deficiency, to demonstrate the ability to achieve a target AUC range, to establish that PK-guided 5-FU dosing decreases the incidence of 5-FU related toxicities, to establish the sensitivity, specificity and predictive values of the DPYD genotyping test and to optimize the sampling moment of 5-FU in order to minimize patient discomfort related to TDM procedures

Study design:

The study is designed as a single-centre prospective inception cohort study. All patients will be screened for DPD deficiency by DPYD genotyping and separated into two groups; DPYD common variants and control group. Patients with DPYD wild-type but who experience CTC grade 3-4 toxicity will also be included in this study as a toxicity group. Patients will be tested with an oral ULT to identify their DPD phenotype and measured an endogenous U/DHU ratio. Therapeutic drug monitoring will be performed to follow-up patients' 5-FU plasma concentration after start chemotherapy treatment. 5-FU plasma concentrations will be monitored until a steady state AUC of 20-30 mg.h/L is reached or maximum 4 treatment cycles is reached.

Study population:

All gastrointestinal cancer patients aged 18 years and older who are scheduled to receive treatment with fluoropyrimidine based chemotherapy.

Treatment:

All patients will be treated with a standard chemotherapy regimen for their respective gastrointestinal cancer. Only 5-FU based regimens will be considered for this study. Patients will receive adjusted 5-FU doses based on their condition, including body surface area, gene activity score or DPD status, and steady state AUC from the previous dose, until their AUC reaches a target range. Patients will continue to receive regular treatment, as long as needed and/or tolerated.

Main study parameters:

The primary outcome of the study is the clearance of 5-FU at steady state (Clss) measured in ml/min. Among cancer patients treated with 5-FU, we will compare the variation in clearance between the four common DPYD variant allele carriers and DPYD wild-type carriers. The secondary study parameters are the incidence of 5-FU related toxicities, U/DHU ratio, DPD phenotype (EM, IM, and PM), 5-FU doses, dosage adjustment and time to reach target AUC (cycle number).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and older
* histological proof of gastro-intestinal cancer
* patient is considered for treatment with capecitabine or 5-FU
* acceptable safety laboratory values
* ECOG performance status 0-2
* able and willing to give written informed consent
* able and willing to undergo blood sampling for DPYD genotyping, DPD phenotyping and pharmacokinetic analysis

Exclusion Criteria:

* symptomatic or uncontrolled central nervous system metastases
* patient who cannot submit itself to the formal follow-up for psychological, social, family or geographical reasons
* women who are pregnant or breast-feeding
* women not consenting to use adequate contraceptive precautions during the study
* significant serious pathology or any instable medical condition (cardiac pathology uncontrolled, myocardial infarction within 6 months before enrolment, systemic active uncontrolled infection, cirrhosis (Child-Pugh score C), renal failure (GFR < 20 ml/min))
* any investigational agent within 4 weeks before enrolment
* cimetidine or sorivudine use (due to drug-drug interactions with 5-fluorouracil and capecitabine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
5-Fluorouracil pharmacokinetics | From enrollment to the end of treatment cycle 4 (the length of each cycle is 14 days)
  The primary objective of this study is to investigate the clearance of 5-FU at steady state (Clss) for the 4 most common DPYD gene variants, compared to the clearance of 5-FU at steady state (Clss) in DPYD wild-type patients and the clearance of 5-FU at steady state (Clss) in assumed DPYD wild-type patients with early grade 3-4 toxicity in order to better define a safe starting dose for 5-FU in DPD deficient patients.

SECONDARY OUTCOMES:
5-FU dose needed to reach target AUC | From enrollment to the end of treatment cycle 4 (the length of each cycle is 14 days)
  The absolute 5-FU dose in mg, needed to reach a target AUC of 20-30 mg.h/L The dose range in each DPYD subgroup will be determined
DPD phenotyping result | From enrollment to the end of treatment cycle 4 (the length of each cycle is 14 days)
  The extent of DPD deficiency as measured by the uracil/dihydrouracil (U/DHU) ratio after oral intake of 1000mg uracil (uracil loading test). A ratio above the threshold value of 2.4 is considered as DPD deficient.
  The range of U/DHU ratio's will be determined for each DPYD subgroup.
Safety and tolerability | From enrollment to the end of treatment cycle 4 (the length of each cycle is 14 days)
  The safety and tolerability of a reduced starting dose of 5-FU in gastrointestinal cancer patients with DPD deficiency as measured by CTC-AE v5 toxicity grading.
  The number of patients in each DPYD subgroup with CTC-AE grade 3 or higher will be determined.
Number of cycles to reach target AUC | From enrollment to the end of treatment cycle 4 (the length of each cycle is 14 days)
  The number of cycles needed to achieve a target AUC range of 20-30 mg.h/L after an adjusted 5-FU dose
Sensitivity, specificity and predictive value of DPYD genotyping | From enrollment to the end of treatment cycle 4 (the length of each cycle is 14 days)
  Calculation of the sensitivity, specificity and predictive values of the DPYD genotyping test, based on both the incidence of unexpected CTC-AE toxicity > grade 3 and the detection of rare DPYD variants detected with DNA sequencing in wild type genotyped patients.
Optimization of 5-FU blood sampling | From enrollment to the end of treatment cycle 4 (the length of each cycle is 14 days)
  Estimation of the most convenient sampling moment (in hours) after start of 5-FU continuous infusion, in order to minimize patient discomfort related to TDM procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Isala Hospital Zwolle, Zwolle, Netherlands

IPD SHARING:
Plan to Share IPD: No
The trial is performed single center at Isala